CLINICAL TRIAL: NCT03911622
Title: Role of Magnetic Resonance Imaging in Evaluation of Uterine Cesarean Section Scar Niche
Brief Title: Mri in Evaluation of Cesarean Section Scar Niche
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kero Wagdy, resident doctor, Assiut University
Other Study IDs: MRI in cesarean scar defects
Record Dates: First submitted 2019-04-07; First posted 2019-04-11 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Cesarean Section; Dehiscence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — medical device that is used as an imaging tool for soft tissues

SUMMARY:
To evaluate cesarean section scar and the lower uterine segment in non pregnant woman by MRI to :

1. Assess the clinical symptoms like postmenstrual spotting or prolonged menstrual bleeding, dysmenorrhea, chronic pelvic pain and dyspareunia and its relation to the presence of cesarean scar defects and its characteristics .
2. development of scoring system and correlating it with the symptoms .

DETAILED DESCRIPTION:
With increasing cesarean section rate nowadays, the risks of cesarean scar defect (CSD) should increase. CSD is defined by ultrasound imaging as a triangular hypoechoic defect in the myometrium at the site of the previous cesarean section scar. However, patients with CSD are sometimes asymptomatic. Yet, some patients with CSD can have symptoms of abnormal uterine bleeding, pelvic pain, infertility, uterine rupture, and potential risks of adverse pregnancy outcome .There is an association between the size of a niche and postmenstrual spotting. women with a history of CS, the depth and shape of the niche were not significant factors, while a larger niche volume was described in women with postmenstrual spotting. in women with gynecological symptoms, the niches were significantly wider in women with postmenstrual spotting, dysmenorrhea or chronic pelvic pain, and the prevalence of postmenstrual spotting or prolonged menstrual bleeding was higher with a larger diameter of the niche .Magnetic resonance imaging (MRI) has recently shown a promise tool for evaluation of uterine scar thickness. As opposed to ultrasonography (USG), which is the current gold standard for this purpose, MRI reduces observer dependence and has a superior multiplanar capability.

MRI can be used for assessment of lower uterine segment. It provides accurate tissue characterization, independent of patient body mass index .

ELIGIBILITY:
Inclusion Criteria:

1. previous lower uterine segment cesarean section before .
2. At least 6 months after the last cesarean section .
3. still regularly menstruating .
4. Absence of other gynecological disease or intrauterine lesions like endometriosis , uterine fibroid .

Exclusion Criteria:

1. Post menopausal women .
2. hysterectomy .
3. Presence of other gynecological disease like endometriosis , uterine fibroids .
4. any general contraindication to MRI as presence of any paramagnetic substance as pacemakers or in severely ill patients or those with claustrophobia, arrhythmic patients .
5. intrauterine devices .
6. bleeding tendency.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients attending at out patient clinic complaining from abnormal bleat gynecology department at Assiut university hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-30 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
MRI pelvis examination (sagittal T2WI ) using 1.5 tesla system Torso phased-array body coil with the patient in the supine position and a moderately full urinary bladder | baseline
  * Pre-designated standard protocols were followed consisting of T1-weighted (T1W) and T2-weighted (T2W) imaging sequences in axial and sagittal planes remaining perpendicular to the long axis of the scar
  * The scar site will be identified as the thinnest portion of LUS and having the lowest signal intensity on T2W imaging.
MRI pelvis examination (sagittal T2WI ) using 1.5 tesla system Torso phased-array body coil with the patient in the supine position and a moderately full urinary bladder | baseline
  - Scar position will be evaluated using relative distance in mm from inferior boundary of scar to external cervix os, which will be measured by curve distance in mm along the endometrium and cervical inner surface.
MRI pelvis examination (sagittal T2WI ) using 1.5 tesla system Torso phased-array body coil with the patient in the supine position and a moderately full urinary bladder | baseline
  Scar thickness in mm will be calculated at the site of the scar .
MRI pelvis examination (sagittal T2WI ) using 1.5 tesla system Torso phased-array body coil with the patient in the supine position and a moderately full urinary bladder | baseline
  Presence of endometrium adjacent to scar will be recorded
MRI pelvis examination (sagittal T2WI ) using 1.5 tesla system Torso phased-array body coil with the patient in the supine position and a moderately full urinary bladder | baseline
  Scar shape were classified as "U" shape, "V" shape and mixed shape, judging from the transitional region from scar to normal uterine or cervical wal

SECONDARY OUTCOMES:
clinical evaluation | baseline
  asking patients about clinical symptoms like postmenstrual spotting , secondary infertility and chronic pelvic pain in order to correlate them with the scar criteria collected by MRI
transabdominal and transvaginal ultrasound examination | baseline
  measuring scar depth in mm .
transabdominal and transvaginal ultrasound examination | baseline
  position in relation to external cervical os and remaining adjacent lower uterine segment
transabdominal and transvaginal ultrasound examination | baseline
  width in mm

CONTACTS AND LOCATIONS:
Overall Officials: Gehan Sayed, PHD, Study Chair — Assiut University; Omran Khodary, MD, Study Director — Assiut University; Hisham Abou Taleb, MD, Study Director — Assiut University

REFERENCES:
- [Background] Jastrow N, Irion O, Roberge S, Bujold E. Clinical importance of appearance of cesarean hysterotomy scar at transvaginal ultrasonography in nonpregnant women. Obstet Gynecol. 2011 Jun;117(6):1438. doi: 10.1097/AOG.0b013e31821e24bc. No abstract available. PMID 21606763
- [Background] Satpathy G, Kumar I, Matah M, Verma A. Comparative accuracy of magnetic resonance morphometry and sonography in assessment of post-cesarean uterine scar. Indian J Radiol Imaging. 2018 Apr-Jun;28(2):169-174. doi: 10.4103/ijri.IJRI_325_17. PMID 30050239
- [Background] Hoffmann J, Stumpp P, Exner M, Grothoff M, Stepan H. Magnetic resonance imaging as additional diagnostic tool in assessment of lower uterine segment in women with previous Cesarean section. Ultrasound Obstet Gynecol. 2019 Feb;53(2):270-272. doi: 10.1002/uog.19046. No abstract available. PMID 29532537
- [Background] Wong WSF, Fung WT. Magnetic Resonance Imaging in the Evaluation of Cesarean Scar Defect. Gynecol Minim Invasive Ther. 2018 Jul-Sep;7(3):104-107. doi: 10.4103/GMIT.GMIT_23_18. Epub 2018 Aug 23. PMID 30254950
- [Background] Gonser M. Re: Prevalence, potential risk factors for development and symptoms related to the presence of uterine niches following Cesarean section: systematic review. Ultrasound Obstet Gynecol. 2014 Sep;44(3):371. doi: 10.1002/uog.14631. No abstract available. PMID 25154489
- [Background] Pomorski M, Fuchs T, Zimmer M. Prediction of uterine dehiscence using ultrasonographic parameters of cesarean section scar in the nonpregnant uterus: a prospective observational study. BMC Pregnancy Childbirth. 2014 Oct 29;14:365. doi: 10.1186/s12884-014-0365-3. PMID 25733122
- [Background] Kumar I, Verma A, Matah M, Satpathy G. Utility of multiparametric MRI in Caesarean section scar characterization and preoperative prediction of scar dehiscence: a prospective study. Acta Radiol. 2017 Jul;58(7):890-896. doi: 10.1177/0284185116675659. Epub 2016 Oct 31. PMID 27799572